CLINICAL TRIAL: NCT07092124
Title: Validation of a Virtual Reality Test for the Assessment of Visually Impaired Patients Undergoing Low Vision Rehabilitation
Acronym: VisionumVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Streetlab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P_VST_2025_2
Record Dates: First submitted 2025-07-11; First posted 2025-07-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test visionumVR (Experimental)
  Interventions: Device: test visionumVR

INTERVENTIONS:
Device: test visionumVR — Two evaluation sessions with VisionumVR one month apart

SUMMARY:
Low vision rehabilitation is a vital part of care for visually impaired patients, who are usually referred to orthoptists to develop visual strategies and optimize residual vision. This rehabilitation significantly improves quality of life by enhancing autonomy and reducing depression. It employs various tools, from traditional exercises to specialized software. Advances in virtual reality (VR) offer new promising opportunities by creating immersive environments tailored to patients' residual vision, increasing motivation and exercise effectiveness. In this context, VisionumVR was developed-a VR test using the Meta Quest 3 headset to assess functional vision during rehabilitation. It evaluates hand-eye coordination, visual discrimination, and visual exploration through a daily-life-inspired task. This standardized 20-minute test aims to measure patients' progress throughout their orthoptic rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient (regardless of visual pathology) who is about to begin or has begun orthoptic low vision rehabilitation;
* Patient requiring at least five orthoptic rehabilitation sessions that can be completed before the end of the study;
* Binocular visual acuity ≥ 1/20 (≤ 1.3 logMAR), regardless of type of vision loss (central, mixed, or peripheral);
* Sufficient knowledge of the French language.

Exclusion Criteria:

* Neurodegenerative diseases or any other condition that could interfere with the planned assessments in this study (known epilepsy and/or history of seizures, dysfunction of the dominant upper limb, etc.);
* Medications that may cause motor, visual, or cognitive impairments (neuroleptics, etc.) or interfere with the study assessments;
* Pregnant women (pregnancy can cause vision fluctuations, and wearing a virtual reality headset is not recommended);
* Participation in another clinical trial that may interfere with the current study;
* Inability to follow instructions or read.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
repetability | Day 0 and Month 1
  Repeatability coefficient of performance on the VisionumVR test

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Régional Basse Vision et Trouble de l'Audition, Angers
  - Institut de Réadaptation Visuelle Saint-Louis, Paris